CLINICAL TRIAL: NCT01795729
Title: Assessment of Revascularization Versus Conservative Treatment in Heart Transplant Patients for a Clinical Event Reduction: THE ARCHER TRIAL
Brief Title: Assessment of Revascularization Versus Conservative Treatment in Heart Transplant Patients for a Clinical Event Reduction
Acronym: ARCHER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081262; 2010-A01516-33 (Other: IDRCB)
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Heart-lung Transplant Rejection
Keywords: Heart transplant; Coronary artery disease; Allograft vascular disease; Coronary stent; Optimal medical therapy; Prognosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Coronary stent+optimal medical therapy (Experimental): Coronary stent on top of optimal medical therapy
  Interventions: Device: Stent; Drug: optimal medical therapy
- 2: Optimal medical therapy (Active Comparator): Optimal medical therapy
  Interventions: Drug: optimal medical therapy

INTERVENTIONS:
Device: Stent — Coronary revascularization
  Other Names: Any type of approved bare metal or drug-eluting coronary stent
  Arms: 1: Coronary stent+optimal medical therapy
Drug: optimal medical therapy — Dual antiplatelet therapy: aspirin and a P2Y12 inhibitor as indicated
  Other Names: Any treatment required at the physicians discretion for the treatment of the patient

SUMMARY:
The aim of the study is to compare optimal medical therapy alone versus percutaneous coronary intervention on top of medical therapy in the setting of heart transplant recipient coronary artery disease in a randomized trial.The primary endpoint assessed at 1 year is the composite of death, myocardial infarction, need for transitory or permanent ventricular assist device implantation, myocardial revascularization, occurrence or worsening of heart failure, any graft dysfunction and/or a decrease of left ventricular ejection fraction of at least 25% compared to baseline. The hypothesis of the study is the superiority of the interventional management over medical therapy alone in preventing the occurrence of the primary endpoint of the study.

DETAILED DESCRIPTION:
The hypothesis of the study is the superiority of the interventional management over medical therapy alone in preventing the occurrence of the primary endpoint of the study assessed 1 year after randomization.

Objectives: To demonstrate the superiority of the interventional management on top of optimal medical therapy over optimal medical therapy alone in preventing the occurrence of the primary endpoint of the study assessed 1 year after randomization

Design : Multicenter, prospective randomized 1 :1, open-label blinded endpoint study

Target population : Heart transplant recipients, aged ≥18 years, without coronary artery disease-related symptoms, with angiographically significant coronary artery stenoses (≥50% anatomically adequate for a revascularization by coronary angioplasty with stent implantation, with no contraindication to dual antiplatelet therapy associating aspirin and a P2Y12 inhibitorfor a duration of 12 monthsand with ni grade IA ACC/AHA indication for revascularization

Inclusion period: 12 months (may be extended based on the inclusion rythme)

Maximum duration of participation for patients : 13 months

Total duration of the study : 37 months

Primary endpoint : The composit of death, myocardial infarction, retransplantation, implantation of transitory or definitve ventricular assist devices, new or worsening heart failure, graft failure and/or a decrease of left ventricular ejection fraction of at least 25% compared to baseline.The occurrence of any event qualifying for the primary endpoint will be assessed by a Cox survival analysis stratified on center.The primary endpoint will be assessed 12 months after randomization.

Secondary endpoints : Any of the individual events defining the primary outcome at 1 year

Number of patients to be included and power calculation : 80 patients per group. A 1 year primary endpoint rate of 30% in the active and 50% in with an inclusion period of 24 months and alpha=5% warants a 90% power using a cox model.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Heart transplant recipient
* Stable clinical situation
* One or several non-critical coronary stenoses (≥ 50% et ≤ 75% visually or QCA-assessed diameter stenosis) considered as adequate for coronary stenting by the operator
* Left ventricular ejection fraction ≥ 40%
* Informed consentement signed by the patient

Exclusion Criteria:

* Acute coronary syndrome
* In-stent restenosis
* Proof of an extensive myocardial ischemia (≥ 7/17 segments ASE model)
* Coronary stenosis considered as critical by the operators with slow flow
* ACC/AHA Class IA indication for revascularization :

  * vessel disease with left ventricular dysfunction
  * Left main stenosis
  * Severe proximal LAD stenosis
* Contra-indication to dual antiplatelet therapy
* Decompensated heart failure at the time of randomization
* Pregnant or breast-feeding women- Patients participating to another clinical research within 30 days before randomization- life expectancy < 1 y
* Patients unable to observe strict medical therapy and follow-up within 1 year after randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The composit of death, myocardial infarction, retransplantation, implantation of transitory or definitive ventricular assist devices, new or worsening heart failure, graft failure and/or a decrease of left ventricular ejection fraction of at least 25% | at 1 year
  The composit of death, myocardial infarction, retransplantation, implantation of transitory or definitive ventricular assist devices, new or worsening heart failure, graft failure and/or a decrease of left ventricular ejection fraction of at least 25% at 1 year

SECONDARY OUTCOMES:
Death at 1 year | at 1 year
myocardial infarction at 1 year | at 1 year
Retransplantation at 1 year | at 1 year
implantation of transitory or definitive ventricular assist devices at 1 year | at 1 year
new or worsening heart failure at 1 year | at 1 year
graft failure and/or a decrease of left ventricular ejection fraction of at least 25% at 1 year compared to baseline | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Farzin BEYGUI, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Pascal LEPRINCE, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris; Saida VARNOUS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié Salpetriere university Hospital - Cardiology, Paris, France